CLINICAL TRIAL: NCT07318623
Title: Comparative Evaluation of Treatment Outcomes Between Damon Ultima and Pitts 21 Pro Bracket Systems; A Randomized Clinical Trial
Brief Title: Comparative Outcomes of Damon Ultima vs Pitts 21 Pro Bracket Systems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hussain Jabar Kadhem, Assistant teacher, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1155425
Record Dates: First submitted 2025-12-30; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Orthodentic Appliances; Orthodontic Pathological Resorption of External Root; Orthodontic Pain; Orthodontic Brackets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Damon ultima bracket group (Active Comparator): Treatment outcome of Damon ultima bracket
  Interventions: Device: Treatment outcome of Damon ultima
- Pitt21 pro bracket group (Active Comparator): Treatment outcome of Pitt21 pro bracket
  Interventions: Device: Treatment outcome of pitt21 pro

INTERVENTIONS:
Device: Treatment outcome of Damon ultima — To compare treatment outcome including duration, root resorption, arch dimension, pain and quality of finishing
  Arms: Damon ultima bracket group
Device: Treatment outcome of pitt21 pro — To compare treatment outcome including duration, root resorption, arch dimension, pain and quality of finishing
  Arms: Pitt21 pro bracket group

SUMMARY:
Title Comparative Evaluation of Treatment Outcomes between Damon Ultima and Pitts 21 Pro Bracket Systems; A Randomized Clinical Trial Abstract Background: The primary advantages of self-ligation brackets include faster archwire removal and ligation, reduced or eliminated need for chairside assistance, secure archwire engagement, and lower bracket-archwire friction, which collectively contribute to a substantial reduction in resistance to sliding and are theorized to enhance the efficiency of initial tooth alignment. This randomized controlled trial (RCT) will be conducted to assess differences in treatment outcomes with these two different self-ligation bracket systems.

Subjects/Materials and Methods: This randomized clinical trial included 40 participants with full permanent dentition (excluding third molars) exhibiting Angle Class I malocclusion with moderate crowding. Patients who were scheduled to undergo orthodontic treatment were allocated into two groups: Damon Ultima and Pitts 21 Pro. The total treatment duration will be measured in months from the bonding day to the completion of treatment, in addition to the number of visits.

Pre-treatment, post-alignment, and post-treatment records were obtained, including intraoral scans (IOS) for assessing alignment efficiency and arch parameters. Periapical radiographs of the upper and lower incisors were taken before and after treatment to measure the amount of root resorption. Treatment outcomes were evaluated using the American Board of Orthodontics (ABO) grading system. Additionally, pain perception and patient treatment perception were assessed.

DETAILED DESCRIPTION:
Comparative Evaluation of Treatment Outcomes between Damon Ultima and Pitts 21 Pro Bracket Systems:

A Randomized Clinical Trial

A Protocol Submitted to the Council of the College of Dentistry, University of Baghdad in Partial Fulfillment of Requirements for the Degree of Doctor of Philosophy in Orthodontics By Hussain Jabar Kadhem B.D.S., M.Sc. (Orthodontics)

Supervised by:

Professor Dr. Mohammed Nahidh B.D.S, M.Sc., Ph.D. (Orthodontics)

Introduction Self-ligating brackets eliminate the need for elastic or wire ligatures by utilizing an integrated opening-and-closing mechanism that holds the archwire in place. Their primary advantages include faster archwire removal and ligation, reduced or eliminated need for chairside assistance, secure archwire engagement, and lower bracket-archwire friction, which collectively contribute to a substantial reduction in resistance to sliding and are theorized to enhance the efficiency of initial tooth alignment .

Previous retrospective studies have shown that the use of self-ligating brackets can reduce treatment times by 4 to 6 months and by 4 to 7 visits when compared with conventional brackets . However, these studies are prone to bias, such as selection, outcome, and recall bias, and confounders.

Although improved treatment efficiency is highly desirable, it has not been a universal finding, particularly for initial alignment and space closure. Some studies have found no difference in the rate of initial alignment with either conventional or self-ligating brackets and have usually compared passive self-ligating brackets with conventional brackets .

Some self-ligating brackets designs can be bulkier, and the sliding mechanism may be prone to binding or breakage, requiring careful clinical management. The claimed clinical superiority, particularly regarding treatment duration, remains a contentious point within the orthodontic literature .

Self-ligating brackets are categorized into two main types: Passive systems, where the clip does not actively exert force on the archwire (e.g., Damon), and Active systems, where the closing mechanism acts as a spring to engage the archwire (e.g., In-Ovation). The choice between systems depends on the desired level of force and control .

Two modern passive self ligating systems are available now namely; Damon Ultima from Ormco, USA and Pitts 21 Pro from OC Orthodontics, USA.

Damon claimed that this system is the first true full expression orthodontic system designed for faster and more precise finishing. Its revolutionary design allows for precise control of rotation, angulation, and torque. The round-sided rectangular Damon Ultima archwire engagement at the horizontal contact points delivers earlier rotation control. Angulation is resolved earlier with vertical contacts, while the engagement at vertical contact points delivers torque control and full expression of the prescription with lighter forces.

On the other hand; Pitts 21 system uses a progressive variation in slot dimensions, transitioning from a square slot (0.021" × 0.021") in the anterior region to a rectangular slot in the posterior portion of the arch-0.021" × 0.023" for premolars and 0.021" × 0.024" for molars. The system claims that this early control of the anterior teeth, achieved through the "Engage Early" wire, allows fuller engagement as early as the second or third appointment without the higher force levels typically associated with large cross-section rectangular archwires, while still providing increased freedom of movement for the posterior teeth .

Finite element analysis comparing Damon Q (rectangular slot) and Pitts 21 (square slot) found that torque moment values, torque expression and Von Mises stress were higher in Pitts 21 brackets at all incisal inclinations .

The systematic review demonstrated that self-ligating brackets do not provide any clinically meaningful reduction in either overall treatment duration or the number of patient visits when compared with conventional bracket systems. Also, most clinical trials comparing self ligating brackets with conventional ligated systems have shown no significant differences in treatment duration, number of appointments or treatment outcomes . Pain perception during initial alignment appears similar between different passive self ligating systems; in a randomized trial comparing Smart Clip and Damon Q, with pain peaked in the first two days . External apical root resorption after treatment with Damon brackets was comparable to conventional brackets .

Comparisons between Damon Ultima and Pitts 21 brackets have not been reported in the literature. Both systems differ in slot geometry and prescribed archwires, which may influence torque, alignment efficiency and arch development. This randomized controlled trial (RCT) will be conducted to assess differences in treatment outcomes with these two bracket systems.

Aim and Objectives Aim The aim of this study will to compare the treatment outcomes of Damon Ultima and Pitts 21 Pro bracket systems.

Primary objective To compare the total treatment time between Damon Ultima and Pitts 21 Pro bracket systems from the day of bracket bonding to the day of debonding.

Secondary objectives

1. Comparing alignment efficiency (measured by Little's irregularity index reduction rate) after each visit between Damon Ultima and Pitts 21 Pro bracket systems and the time taken to reach a well-aligned dental arch.
2. Comparison of pain perception: Patient-reported pain scores will be assessed during the first week following bracket bonding and after first rectangular wire using a 10-cm Visual Analogue Scale (VAS).
3. To compare the amount of orthodontically induced inflammatory root resorption (OIIRR) in the apical region of maxillary and mandibular incisors at start of treatment and at finishing.
4. Evaluating the dental arch dimensions: Measure arch length and widths (inter-canine, inter premolar and inter-molar widths) on digital models before treatment, after leveling/alignment, and at debonding.
5. Recording bracket debonding events and compare failure rates between systems.
6. Evaluating the quality of finished cases using the American Board of Orthodontics - Objective Grading System (ABO-OGS) to grade digital model.

The null hypothesis The null hypothesis I There is no significant difference in treatment duration between patients treated with Damon Ultima brackets and those treated with Pitts 21 Pro brackets.

The null hypothesis II There is no significant difference in alignment efficiency between Damon Ultima and Pitts 21 Pro bracket systems.

The null hypothesis III There is no significant difference in pain perception during treatment between Damon Ultima and Pitts 21 Pro brackets.

The null hypothesis IV There is no significant difference in the amount of external apical root resorption between Damon Ultima and Pitts 21 Pro bracket systems.

The null hypothesis V There is no significant difference in changes in dental arch dimensions between Damon Ultima and Pitts 21 Pro brackets.

The null hypothesis VI There is no significant difference in bracket failure rate between Damon Ultima and Pitts 21 Pro bracket systems.

The null hypothesis VII:

There is no significant difference in bracket failure rate between Damon Ultima and Pitts 21 Pro bracket systems.

Methodology Study design A multi centers, prospective, parallel groups randomized clinical trial with equal allocation to Damon Ultima and Pitts 21 pro systems. The trial will follow CONSORT guidelines for reporting (Figure 1).

Setting This study will be conducted in the orthodontic clinic in the College of Dentistry/ University of, as well as in governmental and private orthodontic centers.

Sample size The sample size was calculated with an alpha level of 5% and 80% power to detect a difference of 3 months in the total duration of treatment, according to the previous data . This revealed that 18 patients in each trial arm would be sufficient to detect this clinical difference (totals 36 patients). In order to account for 10% of dropouts, a total of 40 patients was decided to be collected.

Randomization Participants will be randomly assigned (1:1) to Damon Ultima or Pitts 21 pro using computer generated random blocks of varying sizes (prepared by an independent statistician). Allocation will be concealed in sealed opaque envelopes.

Blinding Operator blinding is not feasible due to the visibly different bracket designs. However, the examiners responsible for assessing outcomes will be blinded to group allocation. This will be achieved by concealing patient names and replacing them with coded numbers, ensuring that the examiner remains unaware of the treatment group.

Intervention procedures The same bonding protocol was applied for all patients, using identical bonding materials (Ormco Enlight Bonding System with Ortho Solo as the primer/bonding agent and 37% phosphoric acid etching gel [FGM, Florida, USA]). Etching was performed for 20 seconds, and curing was carried out using a light-curing unit (Woodpecker, Guilin, China). Smile Arc Protection (SAP) was followed, with minor modifications according to individual case requirements.

Damon Ultima group: Teeth will be bonded with Damon Ultima bracket system. Archwire sequence will be: 0.014 inch CuNiTi, 0.018-inch CuNiTi, 0.014×0.0275-inch CuNiTi and 0.018×0.0275-inch CuNiTi archwires, and 0.019×0.0275-inch stainless steel Ultima finishing archwires.

Pitts 21 Pro group: Teeth will be bonded with Pitts 21 Pro bracket system. Archwire sequence: 0.014-inch thermally Activated NiTi, 0.018 × 0.018-inch thermally Activated NiTi, 0.020×0.020-inch Thermally Activated NiTi, and 0.019 × 0.019-inch stainless steel.

Clinical management Appointment intervals will be scheduled every 8 weeks. Treatment mechanics, including use of inter-arch elastics, bite raiser, and finishing procedures will be standardized. All patients will receive oral hygiene instructions at each visit. In case of bracket failure, brackets will be rebonded using the same system within 3 days, otherwise the case would be considered as dropout.

The case considers as finish if achieve optimal functional occlusion, stable tooth positions, and high-quality esthetics at the end of treatment. Key criteria include establishing Class I molar and canine relationships, normal overjet and overbite, and well-distributed bilateral occlusal contacts without interferences.

Final alignment should show no rotations or spacing, leveled marginal ridges, proper buccolingual inclination, coordinated arch forms, corrected midlines, and a leveled curve of Spee. Esthetic requirements include a consonant smile arc, harmonious tooth proportions, appropriate incisor display, and symmetrical gingival contours.

Outcome measurements and data collection Total treatment duration: It will be measured in months from bonding day to the end of treatment in addition to number of visits.

Alignment efficiency: Little's irregularity index will be measured on 3D digital models at baseline and after completing alignment.

Root resorption: Periapical radiographs of upper and lower incisors before and at end of treatment. EARR will be measure in millimeters on periapical radiographs. Magnification will be corrected based on difference between length of clinical crown and length of crown in periapical radiographs.

Pain perception: 10 cm VAS administered at 24h, 3 days and 5 days after bonding and after first rectangular wire.

Arch dimensions: Including inter-canine, inter-premolar, and inter-molar widths at the buccal cusp tips, as well as arch length, will be measured on digital models at baseline and at the end of treatment. The widths will be measured as the linear distances between the cusp tips of the canines, the buccal cusps of the first premolars, and the mesiobuccal cusps of the first molars. Arch length will be determined as the vertical distance between the midpoint of the two central incisors and the line connecting the mesiobuccal cusp tips of the first molars .

Bracket failure: This will be recorded for any bracket debonding events and tooth location at each visit. Calculate failure rate per bracket and per patient throughout treatment. In case of bracket failure, the same bracket will be treated with sandblast to remove excess composite and re-bond within 3 days.

Quality of finished cases: American Board of Orthodontics - Objective Grading System (ABO-OGS) is used to grade digital model.

Data management and statistical analysis Data will be entered into a secure database with anonymized identifiers. Normality will be tested using the Shapiro-Wilk test. Continuous variables will be summarized as means ± SD or medians with interquartile ranges. Between group comparisons will use independent samples t tests or Mann-Whitney tests as appropriate. Alignment efficiency dental arch dimensions will be analyzed using dependent, independent t-tests and repeated measure ANOVA test. Categorical data (e.g., bracket failure) will be compared using Chi square tests or Fisher's exact tests. A p value < 0.05 will be considered statistically significant.

Data Collection

The following data will be collected and measured during this trial for both groups:

T0: Patients records including full intraoral and extraoral photograph, baseline readings for irregularity index, intraoral scanning, arch dimension measurements on 3 D digital model, radiographs (PA and OPG), oral hygiene instruction and placement of fixed appliances with first archwire.

T1: Complete alignment (measurement of alignment of upper and lower anterior teeth using LII).

T2: At debonding (arch dimension measurement and OIIRR). Pain perception measurement after bracket bonding and after first rectangular wire using visual analog scale (0-10) at 24 hours, 3rd day and 5th day. The number of brackets debonding will be assessed and record each visit.

Stopping Roles If there will be a severe pain in one group that cannot be tolerated by the participants, the study should be terminated.

Budget and Funding The study is self-funded. Ethical Approval The protocol will be submitted to ethics committee. Further Considerations Pilot study: A pilot study will NOT be conducted. Dissemination: Postgraduate Thesis.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of full permanent dentition except the third molars.
2. Class I with moderate crowding requiring fixed appliance therapy and don't need extraction.
3. Good dental hygiene and periodontal health.
4. Good general health; no systemic conditions affecting bone metabolism or pain perception.
5. Normal crown size and shape.
6. No prior orthodontic treatment.
7. Patient has a normal level of vitamin D3 in testing (Vit D3 serum level should be >30).

Exclusion Criteria:

* Severe skeletal discrepancies requiring orthognathic surgery, craniofacial anomalies). Patients with active periodontal disease or medically compromised patients.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To compare the total treatment time between Damon Ultima and Pitts 21 Pro bracket systems. | 24 month
  To compare the total treatment time between Damon Ultima and Pitts 21 Pro bracket systems from the day of bracket bonding to the day of debonding.

SECONDARY OUTCOMES:
Alignment efficiency | up to 6 month
  1. Comparing alignment efficiency (measured by Little's irregularity index reduction rate) after each visit between Damon Ultima and Pitts 21 Pro bracket systems and the time taken to reach a well-aligned dental arch.
2. Comparison of pain perception | through study completion, an average of 2 year
  Patient-reported pain scores will be assessed during the first week following bracket bonding and after first rectangular wire using a 10-cm Visual Analogue Scale (VAS) between Damon Ultima and Pitts 21 Pro bracket systems
the amount of orthodontically induced inflammatory root resorption (OIIRR) | through study completion, an average of 2 year
  compare the amount of orthodontically induced inflammatory root resorption (OIIRR) in the apical region of maxillary and mandibular incisors at start of treatment and at finishing.
Evaluating the dental arch dimensions | through study completion, an average of 2 year
  Measure arch length and widths (inter-canine, inter premolar and inter-molar widths) on digital models before treatment, after leveling/alignment, and at debonding.
bracket debonding events | through study completion, an average of 2 year
  5. Recording bracket debonding events and compare failure rates between systems.
6. Evaluating the quality of finished case. | through study completion, an average of 2 year
  6. Evaluating the quality of finished cases using the American Board of Orthodontics - Objective Grading System (ABO-OGS) to grade digital model.

CONTACTS AND LOCATIONS:
Overall Officials: Hussain Jabar, Principal Investigator — University of Baghdad
Locations (1):
- Collage of dentistry College of Dentistry/ University of Baghdad, Baghdad, Iraq